CLINICAL TRIAL: NCT07089914
Title: Health Surveillance at University of Applied Science Hamburg (HAW) in the Year 2025 to Assess Employees Health and Wellbeing
Brief Title: Health Surveillance at University of Applied Science Hamburg (HAW)
Acronym: HAW-HS 2025
Status: Active, not recruiting | Type: Observational
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: Hamburg University of Applied Sciences/Hochschule für Angewandte Wissenschaften Hamburg (HAW Hamburg) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-02_A
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Social Isolation or Loneliness; Anxiety; Anxiety Acute; Anxiety Depression; Health Behavior; Health Behavior Change; Observational Study; Working Adults; Conditions Influencing Health Status; Anxiety Depression (Mild or Not Persistent); Social Isolation
Keywords: Healthy employees; Health literacy; Disability; Age; Gender; work characteristics; PHQ-4; Self-efficacy; Satisfaction with Life Scale (SWLS); Subjective health status; Job satisfaction; UCLA-LS; HEI-Stress
MeSH Terms: conditions — Social Isolation; Anxiety Disorders; Health Behavior; Lymphoma, Follicular; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- employees: employees at University of Applied Science

SUMMARY:
The aim of Health Surveillance 2025 is to analyze and describe the state of health of employees at University of Applied Science Hamburg, key influencing factors and individual resources.

DETAILED DESCRIPTION:
The aim of Health Surveillance 2025 is to analyze and describe the state of health of students at University of Applied Science Hamburg (HAW), key influencing factors and individual resources. In areas where there is a need for action, the Health Surveillance can provide detailed insights and/or in-depth analyses. The Health Surveillance thus provides information on health-related topics and delivers scientifically sound information as a basis for health-promoting discussions in the subsequent follow-up process at various levels (e.g. faculties). In addition, the Health Surveillance 2025 at University of Applied Science Hamburg contributes to comparability with surveys at other German universities through the use of validated and standardized measuring instruments.

Main hypotheses are

1. The Health Surveillance 2025 gives insights into state of health of employess at HAW, key influencing factors and individual resources.
2. With the Health Surveillance 2025 the health-promotion at HAW can be guided and promotion of mental health (including the reduction of loneliness and discrimination) can be strengthened.
3. The health of employees, their perceived loneliness and discrimination/minorization (disadvantage) interrelates with participation in health promoting activities?
4. Recommendations can be derived for qualification and skills training of multipliers for health-promoting behavior (e.g., MHFA-peers)?

ELIGIBILITY:
Inclusion Criteria:

* German language skills
* Reading and writing skills
* Internet access
* Employee status
* Consent to participate in the study

Exclusion Criteria:

* Illiteracy
* Massively limited cognitive abilities i.e. linguistic components of the digital offerings must be able to be used, and questionnaires completed, or interviews participated in)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All University of Applied Sciences Hamburg employees who wish to take part in the study will be included. Inclusion criteria are germanEnglish language, reading and writing skills, internet access and employee status. Before the start of the survey period and directly before the start of the online survey, all participants will receive all relevant study information and actively declare their consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health literacy | baseline
  10 Items (Lenartz, Söllner & Rudinger, 2014), Range 1 (does not apply/trifft überhaupt nicht zu) - 4 (does fully apply/trifft genau zu), higher scores mean a better outcome
Loneliness | Baseline
  University of California Los Angelese Loneliness Scale (UCLA-LS) - 3 Items (Schobin, Arriagada & Gibson-Kunze, 2024), Range 1 (never/nie) - 5 (very often/sehr oft), higher scores mean a worse outcome

SECONDARY OUTCOMES:
Depression and anxiety | baseline
  Patient Health Questionnaire (PHQ-4) - 4 Items (Kroenke, Spitzer, Williams & Löwe, 2009), Range 0 (not at all/überhaupt nicht) - 3 (nearly every day/beinahe jeden Tag), higher scores mean worse outcome
Subjective health status | baseline
  1 Item (WHO, 1996); Range 1 (very good/sehr gut) - 5 (very poor/schlecht), higher score means worse outcome
Job satisfaction | baseline
  Student satisfaction - 4 Items (Westermann, Heise, Spies & Trautwein, 1996), Range 0 (not at all satisfied/gar nicht zufrieden) - 100 (completely satisfied/vollkommen zufrieden), higher scores mean better outcome
HEI-Stress | baseline
  Higher Education Institution Stress (HEI-Stress) - 3 Items (Schmidt, Sieverding, Scheiter & Obergfell, 2013), Range 0 (not at all stressed/gar nicht gestresst) - 100 (very stressed/sehr gestresst), higher scores mean worse outcome
Self-efficacy | baseline
  5 Items (Jerusalem & Schwarzer, 1999), Range 1 (not at all true/ stimmt nicht) - 4 (exacty true/ stimmt genau) higher scores mean better outcome
Health behaviour | baseline
  3 Items (Burian, Lehnchen, Deptolla, Heinrichs & Stock, 2023) - Range 0 (0 day/ 0 Tage) - 6 (7 days/ 7 Tage) & 1 (I don't eat any fruits or vegetables/ Ich esse keine Früchte oder Gemüse) - 4 (5 portions or more/ 5 Portionen oder mehr) - higher scores mean better outcome
University in transition | baseline
  7 Items (Burian, Lehnchen, Deptolla, Heinrichs & Stock, 2023) - Range 1 (exactly true/ trifft sehr zu) - 4 (not at all true/ trifft überhaupt nicht zu) - higher scores mean worse outcome

OTHER OUTCOMES:
Discriminiation | baseline
  1 Item (SOEP-IS Group, 2022) Range 1 (yes/ ja) - 2 (no/ nein) & 1 Item (DZHW, 2022) multiple choice
Corporate Culture (MOLA) | baseline
  20 Items (Unfallkasse Bahn Bund) - Range 1 (not at all true/ trifft überhaupt nicht zu) - 4 (exactly true/ trifft sehr zu) - higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Principal Investigator — Constructor University Bremen gGmbH & HAW Hamburg
Locations (1):
- Hamburg University of Applied Sciences/Hochschule für Angewandte Wissenschaften Hamburg (HAW Hamburg), Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Due to data security regulations and the approved Data protection concept, sharing is not permitted by the authorities

REFERENCES:
- See also: Description World Health Organization (WHO) (Hrsg.). (2996). Health interview survey: Towards international harmonization of methods and instruments. World He — https://iris.who.int/bitstream/handle/10665/107328/9789289013222-eng.pdf?sequence=1&isAllowe...
- See also: Description Burian, J., Lehnchen, J. Deptolla, Z., Heinrichs, K., Stock, C. (2023). Abschlussbericht zum Vorhaben "Studienbedingungen und (psychische) Gesundheit Studierender: Weiterentwicklung und Erprobung des Bielefelder Fragebogens zu Studienbedingun — https://www.dguv.de/projektdatenbank/0460/fp460_fin_abschlussbericht_mu.pdf
- See also: Kroenke, K., Spitzer, R. L., Williams, J. B. W., & Löwe, B. (2009). An Ultra-Brief Screening Scale for Anxiety and Depression: The PHQ-4. Psychosomatics, 50(6), 613-621. — https://www.researchgate.net/publication/40483064_An_Ultra-Brief_Screening_Scale_for_Anxiety_and...
- See also: SOEP-IS Group (2022). SOEP-IS 2020 - Fragebogen für die SOEP-Innovations-Stichprobe. SOEP Survey Papers 1143: Series A - Survey Instruments (Erhebungsinstrumente). Berlin: DIW Berlin/SOEP. — https://www.diw.de/documents/publikationen/73/diw_01.c.844972.de/diw_ssp1143.pdf
- See also: Deutsches Zentrum für Hochschul- und Wissenschaftsforschung GmbH (DZHW) (2021). Die Studierendenbefragung in Deutschland. Grundprogramm Modul A. Hannover: FDZ-DZHW. — https://doi.org/10.21249/DZHW:sid2021-ins1-att1:1.0.0
- See also: Knispel, J., Wittneben, L., Slavchova, V., & Arling, V. (2021). Skala zur Messung der beruflichen Selbstwirksamkeitserwartung (BSW-5-Rev). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). — https://doi.org/10.6102/ZIS303
- See also: MOLA. Fragebogen für sichere und gesunde Arbeit. Menschen. Organisationskultur. Leistung. Arbeitsgestaltung. — https://www.uv-bund-bahn.de/fileadmin/Dokumente/Fachthemen_Prävention_Dokumente/Psychologie/MOLA/220929_INST_MOLA_Fragebogen_neu.pdf